CLINICAL TRIAL: NCT01131312
Title: Randomized Clinical Trial on Clinical Management of ASCUS and LSIL (ALTS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Schiffman, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 999908076; 08-C-N076
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervix; CIN; HPV; Triage; ASCUS/LSIL; Pap Smear; HPV Test
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Computer random assignment to HPV testing (HC2), cytology (ThinPrep), or immediate colposcopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Cytology (Experimental): Referred to colposcopy if cytology is high grade
  Interventions: Device: Thinprep
- Human Papillomavirus (HPV) (Experimental): Referred to colposcopy if cytology is high grade or HPV +
  Interventions: Device: Hybrid capture 2
- Colposcopy (Experimental): All refer to colposcopy
  Interventions: Procedure: Colposcopy

INTERVENTIONS:
Device: Thinprep — Pap test
  Arms: Cytology
Device: Hybrid capture 2 — Human Papillomavirus (HPV) Deoxyribonucleic Acid (DNA) Test
  Arms: Human Papillomavirus (HPV)
Procedure: Colposcopy — Procedure performed by a healthcare practitioner to examine the cervix, vagina, and vulva.
  Arms: Colposcopy

SUMMARY:
Approximately 65 million Pap smears are performed each year in the United States. The vast majority of results are negative (no abnormality identified) but about 5 percent to 8 percent are reported as abnormal. Most low-grade changes regress spontaneously; only a minority of such lesions would progress to a cancer precursor without treatment. However, there is no way to determine morphologically which patients are at risk or progression. Therefore, both high- and low-grade lesions were often managed with colposcopy and directed biopsy.

Epidemiologic, virologic and molecular studies have clearly demonstrated that human papillomavirus (HPV) is the central cause of cervical cancer. The motivation for the Atypical squamous cells of undetermined significance (ASCUS)- Low grade squamous intraepithelial lesion (LSIL) Triage Study (ALTS) trial was to use the information we have gained about the role of HPV to design better treatment and prevention strategies to reduce the burden of cervical cancer and its precursors.

ALTS consisted of three management strategies: (1) immediate colposcopy of all women; (2) repeat cytology with colposcopy only if the results show a high grade lesion; and (3) HPV testing and repeat cytology in combination, with referral to colposcopy if either the HPV test is positive or the cytology shows a high grade lesion. Four Clinical Centers University of Alabama, Birmingham Alabama (AL); Magee-Womens Hospital, Pittsburgh Pennsylvania (PA); University of Oklahoma, Oklahoma City OK; and University of Washington, Seattle Washington (WA) enrolled approximately 5,000 women with recent diagnosis of ASCUS or LSIL. Participants were followed at six month intervals for a total of 2 years.

The ALTS database and ALTS specimens continue to be a valuable research resource in studies of cervical cancer precursors, screening tests, visual assessment of the cervix and investigation of biomarkers.

DETAILED DESCRIPTION:
Approximately 65 million Pap smears are performed each year in the United States. The vast majority of results are negative (no abnormality identified) but about 5 percent to 8 percent are reported as abnormal. Most low-grade changes regress spontaneously; only a minority of such lesions would progress to a cancer precursor without treatment. However, there is no way to determine morphologically which patients are at risk of progression. Therefore, both high- and low-grade lesions were often managed with colposcopy and directed biopsy. It was anticipated that determining alternative management strategies would yield important potential benefits including fewer medical complications from over treatment, reduced patient anxiety associated with referral for cytologic abnormalities, as well as cost savings.

Epidemiologic, virologic and molecular studies have clearly demonstrated that human papillomavirus (HPV) is the central cause of cervical cancer. The motivation for the ALTS trial was to use the information we have gained about the role of HPV to design better treatment and prevention strategies to reduce the burden of cervical cancer and its precursors.

ALTS consisted of three management strategies: (1) immediate colposcopy of all women; (2) repeat cytology with colposcopy only if the results show a high grade lesion; and (3) HPV testing and repeat cytology in combination, with referral to colposcopy if either the HPV test is positive or the cytology shows a high grade lesion. Four Clinical Centers University of Alabama, Birmingham AL; Magee-Womens Hospital, Pittsburgh PA; University of Oklahoma, Oklahoma City OK; and University of Washington, Seattle WA - enrolled approximately 5,000 women with recent diagnosis of ASCUS or LSIL. Participants were followed at six month intervals for a total of 2 years. The main results from ALTS showed that for women with ASCUS cytology, HPV triage was at least as safe as universal immediate colposcopy in the detection of high-grade lesion and would allow approximately half of women to return to routine follow up without additional procedures (colposcopy). No efficient triage strategy was identified for women with LSIL cytology.

The ALTS database and ALTS specimens continue to be a valuable research resource in studies of cervical cancer precursors, screening tests, visual assessment of the cervix and investigation of biomarkers.

ELIGIBILITY:
* Inclusion Criteria:

  * Diagnosis of atypical squamous cells of undetermined significance (ASCUS) or low-grade squamous intraepithelial lesion (LSIL)
  * 18 years or older
  * Able to give informed consent with reasonable likelihood of follow-up

Exclusion Criteria:

* Previous Hysterectomy
* History of excisional or ablative treatment of cervix, such as laser treatment, radiation therapy, cauterization (burning), freezing or surgery such as cone biopsy or loop electrosurgical excision procedure (LEEP).
* Already known to be pregnant
* Already known to be human immunodeficiency virus (HIV) positive (HIV may negatively affect the clinical history of human papillomavirus (HPV), making triage less appropriate.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5060 (Actual)
Dates: Start 2008-02-20 (Actual); Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Schiffman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The only data sharing is in cervical images which are included as a part of a larger IRB approved release to collaborators completing a data sharing agreement that prohibits re-sharing of data images. The images are shared with limited test results, metadata, and age. The images are saved in encrypted files and shared under individual password protection. Images will only be shared with bonafide researchers who are verified and complete a pilot.
Time Frame: Now and indefinitely.
Access Criteria: The images are saved in encrypted files and shared under individual password protection. Images will only be shared with bonafide researchers who are verified and complete a pilot.

REFERENCES:
- [Background] Boshart M, Gissmann L, Ikenberg H, Kleinheinz A, Scheurlen W, zur Hausen H. A new type of papillomavirus DNA, its presence in genital cancer biopsies and in cell lines derived from cervical cancer. EMBO J. 1984 May;3(5):1151-7. doi: 10.1002/j.1460-2075.1984.tb01944.x. PMID 6329740
- [Background] Cox JT, Lorincz AT, Schiffman MH, Sherman ME, Cullen A, Kurman RJ. Human papillomavirus testing by hybrid capture appears to be useful in triaging women with a cytologic diagnosis of atypical squamous cells of undetermined significance. Am J Obstet Gynecol. 1995 Mar;172(3):946-54. doi: 10.1016/0002-9378(95)90026-8. PMID 7892889
- [Background] Dyson N, Howley PM, Munger K, Harlow E. The human papilloma virus-16 E7 oncoprotein is able to bind to the retinoblastoma gene product. Science. 1989 Feb 17;243(4893):934-7. doi: 10.1126/science.2537532.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytology | Human Papillomavirus (HPV) | Colposcopy
Started | 1839 | 1385 | 1836
Completed | 1414 | 1156 | 1485
Not Completed | 425 | 229 | 351
Not completed — Lost to Follow-up | 425 | 229 | 351

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cytology | Human Papillomavirus (HPV) | Colposcopy | Total
Number analyzed (Participants) | 1839 | 1385 | 1836 | 5060
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 103 | 63 | 99 | 265
  Between 18 and 65 years | 1729 | 1313 | 1729 | 4771
  >=65 years | 7 | 9 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.22 (8.73) | 28.28 (9.62) | 27.24 (8.90) | 27.52 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1839 | 1385 | 1836 | 5060
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 65 | 84 | 230
  Not Hispanic or Latino | 1754 | 1317 | 1751 | 4822
  Unknown or Not Reported | 4 | 3 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 41 | 27 | 40 | 108
  Asian | 48 | 57 | 65 | 170
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 559 | 427 | 569 | 1555
  White | 1180 | 865 | 1146 | 3191
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 16 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1839 | 1385 | 1836 | 5060

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cervical Intraepithelial Neoplasia III (CIN III)
Description: A cervical exam, pap test, human papilloma virus (HPV) deoxyribonucleic acid (DNA) test, and/or colposcopy was performed to detect whether or not a participant had CINIII. CINIII is defined as moderate or severe dysplasia or abnormal cells located on the cervix that can lead to cancer.
Time Frame: up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Cytology | Human Papillomavirus (HPV) | Colposcopy
Number analyzed (Participants) | 1839 | 1385 | 1836
percentage of participants | 10.93 | 10.25 | 10.84

2. Secondary Outcome: Percentage of Participants With Cumulative Detection of Clinical Center Histologically Confirmed Cervical Intraepithelial Neoplasia 2 (CIN2) and Above (High Grade Lesion) Over the 2 Years of the Trial.
Description: Cumulative detection of CIN2 and above was assessed by pathologists who reviewed specimens from cervical pelvic exams (i.e. thin prep pap test, Human papillomavirus (HPV) Deoxyribonucleic acid (DNA) test, and/or colposcopy). Pathologists graded the specimens from CIN2 (moderate grade lesion) to CIN3 (high grade lesion).
Time Frame: up to 2 years
Measure: Number; unit: percentage of particpants
Arm/Group | Cytology | Human Papillomavirus (HPV) | Colposcopy
Number analyzed (Participants) | 1839 | 1385 | 1836
percentage of particpants | 16.69 | 18.12 | 20.75

ADVERSE EVENTS:
Time Frame: Adverse events were to be collected up to 2 years.
Arm/Group | Cytology | Human Papillomavirus (HPV) | Colposcopy
All-Cause Mortality (participants affected / at risk) | 0/1839 | 0/1385 | 0/1836
Serious Adverse Events (participants affected / at risk) | 0/1839 | 0/1385 | 0/1836
Other Adverse Events (participants affected / at risk) | 0/1839 | 0/1385 | 0/1836

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No